CLINICAL TRIAL: NCT03960385
Title: Assessing the Effectiveness of Sanofi Pasteur's Dengue Vaccine (Dengvaxia) Against Hospitalization and Symptomatic Infection in the State of Parana - Brazil
Status: Completed | Type: Observational
Sponsor: Albert B. Sabin Vaccine Institute (Other)
Collaborators: Pan American Health Organization (Other); State of Parana/Health Department of Parana (Unknown); Ministry of Health, Brazil (Other Government); Centro de Estudos Augusto Leopoldo Ayrosa Galvão (Unknown)
Responsible Party: Sponsor
Other Study IDs: DNG10042
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Dengue
Keywords: Dengue; Dengvaxia; Parana; Sanofi Pasteur; Vaccine Effectiveness; Maringa; Foz de Iguacu; Paranagua; Brazil
MeSH Terms: conditions — Dengue | interventions — CYD-TDV vaccine; Dengue Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hospitalized and controls: Age-matched case of hospitalized dengue and non-dengue control
  Interventions: Biological: CYD-TDV
- Outpatient and controls: Age-matched dengue case and non-dengue control
  Interventions: Biological: CYD-TDV

INTERVENTIONS:
Biological: CYD-TDV — Dengue vaccine
  Other Names: Dengvaxia®

SUMMARY:
The study seeks to assess the effectiveness of Sanofi Pasteur´s dengue vaccine (Dengvaxia®) according to the age, dose and municipality of residence in five municipalities of Paraná State. Specific objectives include:

* To assess the effectiveness of Dengvaxia® in preventing dengue hospitalization and dengue symptomatic cases.
* To assess the effectiveness of Dengvaxia® in preventing dengue hospitalization and dengue symptomatic cases according in the following age groups 15 to 18 and 19 to 27 years of age in the municipalities of Maringá, Foz de Iguaçu, Londrina, Sarandi and Paranaguá.
* To assess the effectiveness of Dengvaxia® in preventing dengue hospitalization and dengue symptomatic cases in the following age groups 9 to 14 and 28 to 45 years of age in the municipality of Paranaguá.

DETAILED DESCRIPTION:
The effectiveness of Sanofi Pasteur´s dengue vaccine (Dengvaxia®) according to the age will be assessed in five municipalities of Paraná State - Maringá, Foz de Iguaçu, Londrina, Sarandi and Paranaguá. Any health service located in each of the five municipalities may report a suspected dengue case. However, in all five municipalities, there is a large public emergency service, the UPA. There are currently three UPA in Londrina, two in Maringá and Foz do Iguaҫu and one each in Paranaguá and Sarandi. These facilities are responsible for reporting the majority of suspected dengue cases. In Londrina and Maringá, the private health sector also provides emergency care. The implementation of the study protocol adds a collection of a blood sample for PCR to the existing protocol for addressing suspected dengue cases among individuals within the target vaccination age groups.

The study will count on the activities already carried out by teams of epidemiological surveillance of dengue intensifying the identification of the serotype through the laboratory method RT-PCR (Reverse Transcription Polymerase Chain Reaction) in real time. In addition, the investigators will identify hospitals and health units that attend dengue cases for sample collection, to perform real-time RT-PCR and initial processing of the blood samples collected from the controls.

ELIGIBILITY:
Inclusion criteria for cases:

* Individuals living in the municipalities of Sarandi, Paranaguá, Londrina, Maringá or Foz de Iguaçu in the three stages of vaccination
* Individuals with ages ranging from 9 to 44 years for the municipality of Paranaguá and 15 to 27 years for the municipalities of Sarandi, Londrina, Maringá and Foz de Iguaçu
* All participants who are 18 years of age or older sign the informed consent form
* All minors under the age of 18 who sign the consent form and have the consent form signed by a guardian for the minor
* Case with virological isolation of one of the dengue viruses

Case exclusion criteria:

• Those who have been deprived of their liberty (jails, penitentiaries, drug addicts, etc.) within 15 days before the onset of signs and symptoms

Inclusion criteria for controls:

* Individuals without symptoms for dengue in the 15 days prior to the onset of symptoms of the case
* IgM negative for dengue
* Individuals living in the municipalities of Paranaguá, Londrina, Maringá, Sarandi or Foz de Iguaçu in the three stages of vaccination
* Belongs to the same age group as case
* Participants aged between 9 and 44 years for the municipality of Paranaguá
* Participants 15 to 27 years for the municipalities of Maringá, Foz de Iguaçu, Londrina and Sarandi
* Resides in the same neighborhood as the case, study at the same institution as the case or work in the same company as the case for at least 15 days before the onset of the case symptoms
* Participants that are 18 years of age or older and who sign the informed consent form
* All minors under the age of 18 who sign the consent form and have the consent form signed by a guardian for the minor

Ages: 9 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The effectiveness of Sanofi Pasteur´s dengue vaccine (Dengvaxia®) according to age will be assessed in 5 municipalities of Paraná State - Maringá, Foz de Iguaçu, Londrina, Sarandi and Paranaguá. The municipalities were chosen because they are of medium size and have a history of dengue. The first 4 present a historical series of occurrence of dengue since the 1990s, while in Paranaguá the history of the disease is more recent. Any health service located in each of the five municipalities may report a suspected dengue case. In all five municipalities, there is a large public emergency service, the UPA, which is responsible for reporting the majority of suspected dengue cases. In Londrina and Maringá, the private health sector also provides emergency care.
Sampling Method: Probability Sample
Enrollment: 1854 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Dengue symptomatic case | Aug 2017 - March 2020
  Confirmed (by PCR) case of dengue fever

SECONDARY OUTCOMES:
Dengue hospitalization | Aug 2017 - March 2020
  Hospitalization for severe dengue fever

CONTACTS AND LOCATIONS:
Overall Officials: Denise O Garrett, MD, MSc, Study Director — Albert B. Sabin Vaccine Institute
Locations (1):
- Augusto Leopoldo Ayrosa Galvão Study Center, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No